CLINICAL TRIAL: NCT06396221
Title: "Quick-starting" of a New Combined Hormonal Contraceptive Pills, 15 mg Estetrol/3 mg Drospirenone VS 20 mcg Ethinylestradiol/75 mcg Gestodene Focusing on Ovulation Inhibition: A Single-blind, Randomized Controlled, Non-inferiority Trial
Brief Title: "Quick-starting" of a New Combined Hormonal Contraceptive Pills, 15 mg Estetrol/3 mg Drospirenone VS 20 mcg Ethinylestradiol/75 mcg Gestodene Focusing on Ovulation Inhibition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB0839/66
Record Dates: First submitted 2024-04-25; First posted 2024-05-02 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2024-04

CONDITIONS: Ultrasound Finding: Ovulation Inhibition, Ovarian Activities; Cervical Mucus; Serum Hormonal Profile
Keywords: Quick starting contraception; Estetrol 15 mg and Drospirenone 3 mg; Estetrol/Drospirenone; Ovulation inhibition
MeSH Terms: interventions — Estetrol; drospirenone; Ethinyl Estradiol; Gestodene

STUDY DESIGN:
Intervention Model Description: 1. Ethinylestradiol (EE) 20 mcg/Gestodene 75 mcg (21/7) as control group
  2. Estetrol 15 mg/Drospirenone 3 mg (24/4) as intervention group
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Estetrol 15 mg/Drospirenone 3 mg (24/4) (Experimental)
  Interventions: Drug: Estetrol 15 mg/Drospirenone 3 mg (24/4)
- Ethinylestradiol (EE) 20 mcg/Gestodene 75 mcg (21/7) (Active Comparator)
  Interventions: Drug: Ethinylestradiol (EE) 20 mcg/Gestodene 75 mcg (21/7)

INTERVENTIONS:
Drug: Estetrol 15 mg/Drospirenone 3 mg (24/4) — Completing a pack (28 pills) of Estetrol 15 mg/Drospirenone 3 mg (24/4), starting on day 7-9 of menstrual cycle
  Arms: Estetrol 15 mg/Drospirenone 3 mg (24/4)
Drug: Ethinylestradiol (EE) 20 mcg/Gestodene 75 mcg (21/7) — Completing a pack (28 pills) of Ethinylestradiol (EE) 20 mcg/Gestodene 75 mcg (21/7), starting on day 7-9 of menstrual cycle
  Arms: Ethinylestradiol (EE) 20 mcg/Gestodene 75 mcg (21/7)

SUMMARY:
The goal of this clinical trial is to learn if Estetrol/Drospirenone inhibit ovulation in quick-starting method. It will also learn about the safety of Estetrol/Drospirenone. The main questions it aims to answer are:

1. Does Estetrol/Drospirenone inhibit ovulation inferior to Ethinyl estradiol/Gestodene when starting on Day 7-9 of menstrual cycle?
2. What are the impacts of Estetrol/Drospirenone on ovarian activities when starting on Day 7-9 of menstrual cycle?
3. How does the cervical mucus change when starting Estetrol/Drospirenone on Day 7-9 of menstrual cycle?
4. What are the adverse effects when starting Estetrol/Drospirenone on Day 7-9 of menstrual cycle?

Researchers will compare Estetrol/Drospirenone to Ethinyl estradiol/Gestodene to see if Estetrol/Drospirenone inhibit ovulation in quick-starting method.

DETAILED DESCRIPTION:
Participants will:

Take Estetrol/Drospirenone or Ethinyl estradiol/Gestodene starting on day 7-9 of menstrual cycle then every day for 1 pack of the pills.

Visit the clinic on day 1-2, day 7-9, and then every 2-7 days according to ultrasound finding (ovarian activities) until completing of pills to investigate

1. Transvaginal ultrasound
2. Cervical mucus
3. Serum hormonal profiles.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 - 45 years old
2. Body mass index 18-30 kg/m²
3. Menstrual interval within 24 - 38 days
4. Absence of history of estrogen or progestin allergy and Absence of these compatibles with U.S. medical eligibility criteria category 3 - 4
5. Consent to use condom as contraception or have been sterilized

Exclusion Criteria:

1. History of estrogen, progestin or testosterone use within 3 months
2. Current pregnant or within 3 months of breastfeeding
3. Having ovarian cyst(s) or tumor(s)
4. Being a cervical cancer patient or having precancerous cervical lesion

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 36 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Rate of ovulation inhibition and classify ovarian activities using transvaginal ultrasound | 34-36 days
  Visit the clinic on day 1-2, day 7-9, and then every 2-7 days according to ultrasound finding until completing a package of pills
  * Ultrasound will be perform by the researcher (Dr. Sirarat Itthipuripat) using transvaginal probe to all volunteers.
  * To monitor a leading ovarian follicle or follicle-like structures (FLS), that the ultrasound characteristic is the largest hypoechoic part (follicle) among both ovaries, to classify the ovarian activity by modified Hoogland's score (combined the result with hormonal profile: Estradiol, Progesterone) and assess rate of ovulation, that identify from postovulatory image defined as follows:
  * Image observed after abrupt disappearance of FLS or
  * Image observed after reduction in size of the leading follicle > 4 mm at 2 consecutive visits or
  * Hemorrhagic or cystic corpus luteum
  * The detail in measuring the size of an FLS is the average of 3 longest sides perpendicular to each other in millimeter

SECONDARY OUTCOMES:
Level of serum hormonal profiles: Estradiol, Progesterone, LH | Cervical mucus classification
  Visit the clinic on day 1-2, day 7-9, and then every 2-7 days according to ultrasound finding
  * Blood test to measure estrogen level in picogram/milliliter, progesterone level in nanogram/milliliter and LH level in International unit per liter
  * Volunteers will be placed in a 5 ml clot activator tube and sent to the endocrinology laboratory medical operation center within 30 minutes after blood draw.
Cervical mucus | 34-36 days
  Visit the clinic on day 1-2, day 7-9, and then every 2-7 days according to ultrasound finding
  * Using Tuberculin syringe 1 mL to suck cervical mucus from the endocervical canal (1 cm deep from external cervical os)
  * Assess the results of cervical mucus collected immediately according to WHO 2010, consisting of volume (milliliter), viscosity, ferning appearance, Spinnbarkeit (centimeter), and cellularity (cell/high power field), under microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Somsook Santibenchakul, Master, Study Director — Obstetric and gynecology department, Faculty of medicine, Chulalongkorn University
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ittipuripat S, Phutrakool P, Uaamnuichai S, Porntawansak G, Wongwathanavikrom R, Utaipatanacheep P, Santibenchakul S. Delayed start of estetrol drospirenone versus ethinyl estradiol gestodene for ovulation inhibition in a noninferiority randomized controlled trial. Sci Rep. 2025 Dec 12;15(1):43682. doi: 10.1038/s41598-025-27467-y. PMID 41388035